CLINICAL TRIAL: NCT02523378
Title: Edmonton Symptom Assessment Scale: Time Duration of Self-Completion Versus Assisted-Completion in Advanced Cancer Patient: a Randomized Controlled Trial
Brief Title: Edmonton Symptom Assessment Scale: Self-Completion vs. Assisted-Completion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0284; NCI-2015-01441 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Recurrent; Locally advanced; Metastatic; Edmonton Symptom Assessment Scale; ESAS; Survey; Interview; Symptom questionnaire
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESAS Self-Administration - Group A (Experimental): Participants complete the symptom questionnaire alone. It is then counterchecked by health care professional (HCP).
  Interventions: Behavioral: Edmonton Symptom Assessment Scale; Behavioral: Interview
- ESAS Assisted-Completion - Group B (Experimental): Participants complete the symptom questionnaire with the help of the research nurse or assistant.
  Interventions: Behavioral: Edmonton Symptom Assessment Scale; Behavioral: Interview

INTERVENTIONS:
Behavioral: Edmonton Symptom Assessment Scale — Participants complete the symptom survey alone, or with the help of a research nurse or assistant.
  Other Names: Survey; Questionnaire
Behavioral: Interview — After completion of the symptom questionnaire, participants asked if they preferred completing the questionnaire alone, or if they preferred to have a nurse help them answer the questions.

SUMMARY:
The goal of this research study is to learn how easy participants think it is to complete a symptom questionnaire.

DETAILED DESCRIPTION:
If participant agrees to take part in the study, basic information about them will be collected from their medical record (such as their age, gender, ethnicity, religion, diagnosis, marital status, educational level, performance status, and any drugs they may have taken in the past or are currently taking).

Participant will also be given a list of words and asked to read them out loud. The research nurse or assistant will write down if participant pronounced the words correctly. This should take up to 7 minutes.

Participant will then be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If participant is enrolled in Group 1, they will complete the symptom questionnaire alone and then a research nurse or assistant will go over their answers with them.
* If participant is enrolled in Group 2, they will complete the symptom questionnaire with the help of the research nurse or assistant.

After participant has completed the symptom questionnaire, they will be asked if they preferred completing the questionnaire alone or if they preferred to have a nurse help them answer the questions. This should take about 1 minute to answer.

Length of Study:

It should take about 15 minutes total to complete the study. Patient's participation on this study will end after they have completed the symptom questionnaire.

Additional Information:

Participant is taking part in this study alone. Participant's family members will not be in the room with them.

This is an investigational study.

Up to 128 participants will be enrolled in the study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of advanced cancer, including recurrent, locally advanced, or metastatic cancer
2. Patients must know their cancer diagnosis
3. Patients referred for consultation to the Supportive Care team
4. Age >/= 18
5. Patients must be able to understand, read, write, and speak English
6. Patients have never done the ESAS before
7. Patients must sign an informed consent
8. Ability to independently complete the study as assessed by the research staff

Exclusion Criteria:

1. Patients who have clinical evidence of cognitive impairment as determined by the research staff
2. Patients who have already done the ESAS in the past.
3. Patients who are considered to be in severe physical or emotional distress based on the assessment by the research staff
4. Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Time Duration of Self-Completion of Edmonton Symptom Assessment Scale (ESAS) by Advanced Cancer Participants (ACP) vs. Assisted-Completion with a Health Care Professional (HCP) | 1 day
  Two group t-test used with significance level of 5%, a total of 128 patients (64 patients/group) will give 80% power to detect the difference of 1.5 minutes (4 minutes in Group A vs 5.5 minutes in Group B) in overall time, given a common standard deviation of 3, which corresponds to an effect size of 0.5.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org